CLINICAL TRIAL: NCT07390591
Title: Intravesical Gentamicin Coupled With Lactobacillus Rhamnosus for Urinary Health- Early Career
Brief Title: Patient and Caregiver Perspectives on Intravesical Instillations for Urinary Symptoms
Status: Recruiting | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: STUDY00009066; CDMRP-SC230144P1 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs (CDMRP))
Record Dates: First submitted 2025-12-09; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries; Neurogenic Lower Urinary Tract Dysfunction; Neurogenic Bladder
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational qualitative study is to learn about the experiences and perspectives of patients with neurogenic lower urinary tract dysfunction (NLUTD) and their caregivers regarding different types of intravesical instillations used for urinary health. The study aims to understand the perceived benefits, challenges, and opportunities related to Lactobacillus-only, gentamicin-only, and combined gentamicin-Lactobacillus instillations. The main question this study seeks to answer is:

1. Determine patient and caregivers' preferences, and overall experiences regarding intravesical therapeutics for urinary symptoms and UTI

Researchers will compare responses from four groups: participants who have used Lactobacillus-only instillations, gentamicin-only instillations, combined gentamicin-Lactobacillus instillations, and caregivers who have experience supporting instillations.

Participants will take part in a one-hour semi-structured interview and may be contacted for brief follow-up discussions to clarify findings. Interviews will be audio-recorded, transcribed, and analyzed using qualitative data software to identify themes related to treatment preferences and acceptability.

DETAILED DESCRIPTION:
Participants in this study will engage in an in-depth qualitative semi-structured interview process designed to explore their experiences with intravesical instillation practices. Each participant will complete a one-hour interview, during which they will be asked about their personal routines, decision-making factors, and perceptions related to bladder instillations. To ensure accuracy of interpretation, participants may also be invited to take part in brief follow-up discussions lasting no more than 30 minutes each. These follow-up interactions will occur within 12 months of the initial interview, and the total participation time will not exceed 2.5 hours over the study period.

All interviews will be audio-recorded, transcribed, reviewed for accuracy, and analyzed using a secure, cloud-based qualitative data analysis platform that allows linked review of audio and transcript files. Interviews will continue until data saturation is reached, meaning no new concepts emerge from additional participants.

ELIGIBILITY:
Inclusion Criteria:

Criteria for patients:

* Age 18+
* Diagnosis of NLUTD
* Chronic catheter usage (minimum 6 months), either intermittent catheterization or indwelling catheter
* Community-dwelling
* Experience using intravesical Lactobacillus, gentamicin, or combination of the two

Criteria for caregivers:

* Age 18+
* Care for patient with diagnosis of NLUTD
* Care for patient who has used catheters chronically (minimum 6 months)
* Experience facilitating patients' use of intravesical Lactobacillus, gentamicin, or combination of the two

Exclusion Criteria:

* Psychiatric or psychologic conditions impacting ability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from populations that have used Lactobacillus, gentamicin, or combination of the two.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Advancing intravesical instillation for urinary health | 12 months
  Qualitative interviews will be coded, and themes how to advance intravesical instillation for urinary health will emerge.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Valeria Aguirre Guemez, MD, Principal Investigator — MedStar National Rehabilitation Hospital
Locations (1):
- Medstar National Rehabilitation Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No